CLINICAL TRIAL: NCT03835455
Title: A Mixed Methods Study to Determine the Acceptability and Feasibility of Providing Finger Foods as Nutritional Support for Patients After Stroke in Hospital
Brief Title: Acceptability and Feasibility of Finger Foods
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: 40715
Record Dates: First submitted 2019-01-25; First posted 2019-02-08 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Stroke, Acute
Keywords: Finger food
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will investigate the feasibility of using a finger food menu on an acute stroke rehabilitation ward. This study has a mixed methods design, with quantitative, qualitative and economic components which will be used to inform a future randomised control trial.

ELIGIBILITY:
Inclusion Criteria:

* Current patient on stroke rehabilitation ward
* 65 years or older
* Normal textured food

Exclusion Criteria:

* On the end of life pathway
* Partial or full enteral feeding
* Significant food allergies, intolerances or other dietary restrictions that could not be catered for by the finger food menu.
* Unable to give consent or no consultee able to consent on behalf of patient
* In a side room on the ward

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: On stroke rehabilitation ward
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Eligibility rate | 6 months
  Number of patients eligible for study based on inclusion and exclusion criteria
Recruitment rate | 6 months
  Number of patients approached vs number of patients recruited to the study
Attrition rate | 6 months
  Number of participants without fully completed outcome measures

SECONDARY OUTCOMES:
Dietary intake of participants over 3 mealtimes | 3 mealtimes
  Estimation of dietary intake over 3 mealtimes. This will include a standard mealtime and 2 meals when the finger menu is offered. This will be measured as energy and protein intake.
Costs of implementing a finger food menu | 6 months
  A cost consequence analysis will be used to describe direct and indirect costs associated with providing a finger food menu.
Fidelity of intervention | 6 months
  Fidelity determined through observation field notes

OTHER OUTCOMES:
Patient experience | 6 months
  Semi-structured interviews with participants to determine patient experience
Staff experience | 6 months
  Semi-structured interviews with staff to determine facilitators and barriers to using the menu on the ward

CONTACTS AND LOCATIONS:
Overall Officials: Milly Heelan, Principal Investigator — University of Southampton
Locations (1):
- University Hospital Southampton NHS trust, Southampton, United Kingdom